CLINICAL TRIAL: NCT06037629
Title: Premature Enhanced Automated Capture of Comfort Knowledge (PEACOCK)
Brief Title: Premature Enhanced Automated Capture of Comfort Knowledge
Acronym: PEACOCK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Arthur Howard, Principal Investigator, Newcastle University
Other Study IDs: 299441
Record Dates: First submitted 2023-03-29; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain; Pain, Procedural; Agitation; Discomfort
MeSH Terms: conditions — Acute Pain; Pain, Procedural; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm neonates in intensive care: Preterm neonates born <36 completed weeks of gestation with postmenstrual age <36 weeks

SUMMARY:
The goal of this observational study is to develop methods that could provide continual monitoring of comfort levels for preterm neonates in hospitals.

DETAILED DESCRIPTION:
As preterm neonates have not developed ways to communicate how they are feeling like children or adults do, clinicians must rely on their own understanding and professional judgements to decide how comfortable they are. It is known that preterm neonates can display emotion through ways such as facial expressions, body movements and changes in their physiology such as heart rate. The investigators will record both behavioural (audiovisual) and physiologic (heart rate, blood oxygen saturation) signals during routine clinical procedures ranging from comforting, through discomforting to painful that are necessary as part of high-quality medical care.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants born <36 completed weeks of gestation
* Medically stable
* Written informed consent from parents

Exclusion Criteria:

* Infants with significant brain, spine, or congenital abnormality
* Parents unwilling to provide consent
* Infants with postmenstrual age >36 weeks

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates hospitalised in the Royal Victoria Infirmary Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score Before Procedure | 1 minute recording before procedure
  Score provided by nurses from Neonatal Pain, Agitation & Sedation Scale. Pain/Agitation scores range from 0-13, higher scores indicate higher pain/agitation levels.
Audiovisual signal Before Procedure | 1 minute starting before procedure
  Bedside recording using camera and microphone.
Physiologic Signal Before Procedure: Heart Rate | 1 minute starting before procedure
  Heart rate captured by bedside ECG monitor
Physiologic Signal Before Procedure: Blood Oxygen Saturation | 1 minute starting before procedure
  Blood oxygen saturation captured by bedside oximetry monitor
Pain Score During Procedure | 1 minute recording during procedure
  Score provided by nurses from Neonatal Pain, Agitation & Sedation Scale. Pain/Agitation scores range from 0-13, higher scores indicate higher pain/agitation levels.
Audiovisual Signal During Procedure | 1 minute during procedure
  Bedside recording using camera and microphone
Physiologic Signal During Procedure: Heart Rate | 1 minute during procedure
  Heart rate captured by bedside ECG monitor
Physiologic Signal During Procedure: Blood Oxygen Saturation | 1 minute during procedure
  Blood oxygen saturation captured by bedside oximetry monitor
Pain Score After Procedure | 1 minute recording immediately after procedure
  Score provided by nurses from Neonatal Pain, Agitation & Sedation Scale. Pain/Agitation scores range from 0-13, higher scores indicate higher pain/agitation levels.
Audiovisual Signal After Procedure | 1 minute immediately after procedure
  Bedside recording using camera and microphone
Physiologic Signal After Procedure: Heart Rate | 1 minute immediately after procedure
  Heart rate captured by bedside ECG monitor
Physiologic Signal After Procedure: Blood Oxygen Saturation | 1 minute immediately after procedure
  Blood oxygen saturation captured by bedside oximetry monitor

CONTACTS AND LOCATIONS:
Locations (1):
- The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No